CLINICAL TRIAL: NCT00342667
Title: Clinical, Biochemical, Histological and Biophysical Parameters in the Prediction of Cerebral Palsy in Patients With Preterm Labor and Premature Rupture of Membranes
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999997066; OH97-CH-N066
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Preterm Birth; Pregnancy
Keywords: Pregnancy; Pregnancy Complications; Natural History
MeSH Terms: conditions — Premature Birth; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: patients with preterm labor/contractions and preterm premature rupture of membranes

SUMMARY:
A major goal of modern perinatal and neonatal medicine is to reduce the rate of developmental disabilities, especially mental retardation. Cerebral palsy is frequently associated with neurologic abnormalities and mental retardation. Improvements in neonatal intensive care have resulted in improved survival of very low birthweight infants but also in an increased frequency of cerebral palsy. Prematurity is a leading risk factor for cerebral palsy. Two thirds of preterm neonates are born to mothers with preterm labor with intact membranes or preterm premature rupture of membranes. A growing body of evidence suggests that these conditions are heterogeneous. This is an observational cohort study designed to identify the mechanisms of disease in patients with preterm labor/contractions and preterm premature rupture of membranes and to describe the relationship between clinical, biochemical, histological, biophysical parameters and the development of infant neurological disorders.

DETAILED DESCRIPTION:
A major goal of modern perinatal and neonatal medicine is to reduce the rate of developmental disabilities, especially mental retardation. Cerebral palsy is frequently associated with neurologic abnormalities and mental retardation. Improvements in neonatal intensive care have resulted in improved survival of very low birthweight infants but also in an increased frequency of cerebral palsy. Prematurity is a leading risk factor for cerebral palsy. Two thirds of preterm neonates are born to mothers with preterm labor with intact membranes or preterm premature rupture of membranes. A growing body of evidence suggests that these conditions are heterogeneous. This is an observational cohort study designed to identify the mechanisms of disease in patients with preterm labor/contractions and preterm premature rupture of membranes and to describe the relationship between clinical, biochemical, histological, biophysical parameters and the development of infant neurological disorders.

ELIGIBILITY:
* INCLUSION CRITERIA:

Consecutive patients admitted with the diagnosis of preterm labor/contractions or PROM.

"Preterm labor/contractions" will be defined as:

1. gestational age: 20-36 weeks;
2. intact membranes; and
3. regular uterine contractions greater than or equal to 8 in 60 minutes.

Preterm PROM will be defined as:

1. gestational age 20-36 weeks; and
2. spontaneous rupture of membranes as diagnosed by sterile speculum examination confirming pooling of amniotic fluid in the vagina, a positive Nitrazine test result, and a positive ferning test result. In cases of suspected but unconfirmed preterm PROM, indigo carmin instillation will be performed. The vaginal leakage of indigo carmin will confirm the diagnosis in these cases.

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This is an observational cohort study designed to identify the mechanisms of disease in patients with preterm labor/contractions and preterm premature rupture of membranes and to describe the relationship between clinical, biochemical, histological, biophysical parameters and the development of infant neurological disorders.@@@
Sampling Method: Probability Sample
Enrollment: 4673 (Actual)
Dates: Start 1997-12-08 (Actual); Primary Completion 2014-09-15 (Actual); Study Completion 2014-09-15 (Actual)

PRIMARY OUTCOMES:
Establish the relationship between these pathologic sub- groups (i.e., intrauterine infection and non infection associated preterm labor/contractions and preterm PROM ) and short and long term neonatal outcome. | 1. gestational age: 20-36
  Establish the relationship between these pathologic sub- groups (i.e., intrauterine infection and non infection associated preterm labor /contractions and preterm PROM ) and short and long term neonatal outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Romero, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (5):
- United States (2):
  - National Institute of Child Health and Human Development (NICHD), 9000 Rockville, Bethesda, Maryland
  - Hutzel Women's Hospital, Detroit, Michigan
- Sotero del Rio Hospital, Puente Alto, Chile
- Ben Gurion University /Soroka Medical Center, Beersheba, Israel
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Nelson KB, Dambrosia JM, Ting TY, Grether JK. Uncertain value of electronic fetal monitoring in predicting cerebral palsy. N Engl J Med. 1996 Mar 7;334(10):613-8. doi: 10.1056/NEJM199603073341001. PMID 8592523
- [Background] Nicholson A, Alberman E. Cerebral palsy--an increasing contributor to severe mental retardation? Arch Dis Child. 1992 Aug;67(8):1050-5. doi: 10.1136/adc.67.8.1050. PMID 1520012
- [Background] Cummins SK, Nelson KB, Grether JK, Velie EM. Cerebral palsy in four northern California counties, births 1983 through 1985. J Pediatr. 1993 Aug;123(2):230-7. doi: 10.1016/s0022-3476(05)81693-2. PMID 8345418